CLINICAL TRIAL: NCT06656494
Title: A Phase 1 Study of ICP-248 in Combination With Azacitidine for the Treatment in Patients With Myeloid Malignancies.
Brief Title: ICP-248 in Combination With Azacitidine for the Treatment in Patients With Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Beijing InnoCare Pharma Tech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ICP-CL-01205
Record Dates: First submitted 2024-10-21; First posted 2024-10-24 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Acute Myelogenous Leukemia; Myelodysplastic Syndromes (MDS)
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ICP-248 in combination with azacitidine (Experimental)
  Interventions: Drug: ICP-248; Drug: Azacitidine

INTERVENTIONS:
Drug: ICP-248 — Eligible patients will receive ICP-248 orally as per the protocol，once daily for every 28 days as one treatment cycle
Drug: Azacitidine — Eligible patients will receive azacitidine subcutaneously or intravenously as per the protocol，once daily on days 1-7 of each 28-day cycle.

SUMMARY:
Evaluate the safety, tolerability, pharmacokinetics, and preliminary efficacy of ICP-248 in combination with azacitidine in patients with acute myelogenous leukemia and Myelodysplastic Syndromes.

ELIGIBILITY:
Inclusion Criteria:

Eligible subjects must meet all of the following criteria:

1. Subject must have confirmation of diagnosis of AML (except for acute promyelocytic leukemia [APL]) or MDS per 2016 World Health Organization (WHO) criteria.
2. For AML (except for APL) cohort:

   1. Previously treated relapsed/refractory AML subjects
   2. Treatment-naïve AML subjects should be: ≥60 years of age OR ≥18 years and <60 years will be eligible if the subject has at least one of the following co-morbidities, which make the subject unfit for intensive chemotherapy
3. For MDS cohort: Adult TN MDS and R/R MDS: revised International Prognostic Scoring System (IPSS-R) score > 3 and bone marrow blasts ≥ 5%.
4. Subject must have a projected life expectancy of at least 12 weeks.
5. Subject must have adequate renal function as demonstrated by a creatinine clearance ≥ 30 mL/min; determined via urine collection for 24-hour creatinine clearance or by the Cockcroft-Gault formula.
6. Subject must have adequate liver function

Exclusion Criteria:

1. R/R AML or R/R MDS with no response or intolerance to post azacitidine or BCL-2i.
2. Subject has acute promyelocytic leukemia (French-American-British Class M3 AML) .
3. Subject has known central nervous system (CNS) leukemia.
4. Suggest patients with active hepatitis B or C virus infection
5. History of immunodeficiency, including a positive human immunodeficiency virus (HIV) antibody test.
6. Subjects have another active malignancy within the past 2 years before study entry, except for curatively treated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 266 (Estimated)
Dates: Start 2024-12-18 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Incidence, type, and severity of dose-limiting toxicity (DLT). | 2.5 years
Recommended phase II dose (RP2D) and/or maximum tolerated dose (MTD). | 2.5 years
The incidence, nature, and severity of adverse events (AEs) as assessed per National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE v5.0) criteria. | 2.5 years
AML cohort:Composite complete remission rate by Investigator per ELN 2017 criteria. | 2.5 years
AML cohort：Composite complete remission rate by completion of cycle 2 by Investigator per ELN 2017 criteria. | 2.5 years
MDS cohort：mOR rate, including CR, mCR, and PR, assessed by Investigator at any time point during the study per revised IWG 2006 MDS Criteria. | 2.5 years

SECONDARY OUTCOMES:
AML cohort：Composite complete remission rate: The proportion of subjects with complete remission (CR) and CR with incomplete hematologic recovery (CRi) by Investigator per European Leukemia Net (ELN) 2017 criteria. | 2.5 years
AML cohort：Composite complete remission rate by completion of cycle 2 by Investigator per ELN 2017 criteria. | 2.5 years
The incidence, nature, and severity of adverse events (AEs) as assessed per NCI-CTCAE v5.0 criteria. | 2.5 years
Maximum concentration (Cmax)of ICP-248. | 2.5 years
Area under the curve (AUC) of ICP-248. | 2.5 years
Time of maximum observed plasma(Tmax)of ICP-248. | 2.5 years
Trough concentration(Ctrough) of ICP-248. | 2.5 years
Apparent clearance (CL/F) of ICP-248. | 2.5 years
AML cohort：Partial Response (PR) by investigator per ELN 2017 criteria. | 2.5 years
AML cohort：Overall survival (OS) by investigator per ELN 2017 criteria. | 2.5 years
AML cohort：Duration of Response (DOR) by investigator per ELN 2017 criteria. | 2.5 years
AML cohort：Event-free Survival (EFS) by investigator per ELN 2017 criteria. | 2.5 years
AML cohort：Relapse-free Survival (RFS) by investigator per ELN 2017 criteria. | 2.5 years
AML cohort：Morphologic leukemia-free state (MLFS) by investigator per ELN 2017 criteria. | 2.5 years
MDS cohort：Modified overall response (mOR) rate, including CR, marrow complete response (mCR), and PR, assessed by Investigator at any time point during the study per revised International Working Group (IWG) 2006 MDS Criteria | 2.5 years
MDS cohort：Complete remission(CR) rate by Investigator per revised IWG 2006 MDS Criteria | 2.5 years
MDS cohort：Event-free survival (EFS) by Investigator per revised IWG 2006 MDS Criteria | 2.5 years
MDS cohort：Duration of modified overall response (DmOR) by Investigator per revised IWG 2006 MDS Criteria | 2.5 years
MDS cohort：Overall survival(OS) by Investigator per revised IWG 2006 MDS Criteria | 2.5 years
MDS cohort：Marrow complete response (mCR) rate by Investigator per revised IWG 2006 MDS Criteria | 2.5 years

CONTACTS AND LOCATIONS:
Locations (15):
- NYU Langone Health, New York, New York, United States
- China (14):
  - Anhui Provincial Hospita, Hefei, Anhui
  - Peking University People's Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - Guangdong Provincial People's Hospital, Guangzhou, Guangdong
  - Nanfang Hospital Southern Medical University, Guangzhou, Guangdong
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - Shengjing Hospital of China Medical University, Shengyang, Liaoning
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Tianjin People's Hospital, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang